CLINICAL TRIAL: NCT05406765
Title: Spinal Analgesia for Laparoscopic Abdominoperineal Rectal Amputation Using an Enhanced Recovery After Surgery Program: a Randomized Double-blind Placebo-controlled Trial
Brief Title: Enhanced Recovery After Laparoscopic Colorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Project 2805
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-05

CONDITIONS: Rectal Cancer; Postoperative Pain
MeSH Terms: conditions — Rectal Neoplasms; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization, allocation, and blinding: Randomization will be conducted by using sealed, opaque envelopes. An independent colleague at the Clinical Research Department will randomize these envelopes in blocks of 5. These envelopes will be stacked and stored outside the operating room. The upper envelope will be opened by the attending anesthesiologist when an included patient arrives in the operating theater. The patient, surgical team, nurses on the ward, and researcher team will be blinded. Only the attending anesthetic team will be aware of the randomization. They will be instructed not to tell the patient or any other health care worker which group the patient was allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal (Active Comparator): Spinal anesthesia
  Interventions: Drug: Bupivacaine Injection
- Placebo (Placebo Comparator): Placebo spinal
  Interventions: Drug: Bupivacaine Injection

INTERVENTIONS:
Drug: Bupivacaine Injection — One group will receive bupivacaine 15 mg and morphine 100 ug intrathecally
  Other Names: Marcain

SUMMARY:
Investigators would like to test the effects of spinal anesthesia as an adjunct to general anesthesia in patients undergoing laparoscopic abdominoperineal rectal amputation. Investigators hypothesize that spinal anesthesia as an adjunct to general anesthesia will reduce postoperative pain and opioid requirements.

DETAILED DESCRIPTION:
Effective pain management after laparoscopic rectal surgery is a fundamental requirement in an enhanced recovery after surgery program (ERAS). Opioids remain the mainstay for postsurgical pain despite well documented side effects including sedation, dizziness, nausea, vomiting, constipation, physical dependence, tolerance, and respiratory depression. Spinal analgesia as an adjunct to general anesthesia has not been studied in laparoscopic rectal surgery, but data from studies of patients undergoing colon cancer resection indicate a positive analgesic effect of spinal anesthesia as an adjunct to general anesthesia. When an ERAS program was used for laparoscopic colonic resection, It has been showed that an intrathecal mixture of bupivacaine and morphine was associated with less postoperative opioid consumption. In a more recent paper intrathecal morphine was a more effective method for treating postoperative pain in laparoscopic colon surgery than intravenous opioids within an ERAS program. In the present proposal the investigators would like to test the effects of spinal anesthesia as an adjunct to general anesthesia in patients undergoing laparoscopic abdominoperineal rectal amputation. It was hypothesized that spinal anesthesia as an adjunct to general anesthesia would reduce postoperative pain and opioid requirements.

ELIGIBILITY:
Inclusion Criteria

*All patients undergoing laparoscopic abdominoperineal rectal amputation for rectal cancer * Age 18-100 years are eligible for enrollment in the study.

Exclusion Criteria

* ASA IV,
* BMI>35,
* contraindication to spinal analgesia
* allergy to any of the drugs used in this study protocol,
* chronic use of opioids or steroids,
* liver or renal impairment,
* patients scheduled for synchronous laparoscopic liver metastatic surgery
* inability to communicate in Norwegian.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Nummeric rating scale (0-10), where 10 indicate worst possible pain. | 48 hours after surgery
  Worst pain scores in the first 48 hrs.

CONTACTS AND LOCATIONS:
Overall Officials: Lars M Ytrebø, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Antunes M, Baumgartel A, Gjessing PF, Ytrebo LM. Spinal Anaesthesia as an Adjunct to General Anaesthesia for Laparoscopic Abdominoperineal Rectal Amputation. J Pain Res. 2023 May 31;16:1855-1865. doi: 10.2147/JPR.S410019. eCollection 2023. PMID 37284327